CLINICAL TRIAL: NCT06644222
Title: The Effectiveness of Airrosti and TheraBand Exercises on Pain and Disability on Double-Crossed Syndrome in Smart Phone User's Shoulder
Brief Title: Effectiveness of Airrosti and TheraBand Exercises on Double-Crossed Syndrome in Smart Phone User's Shoulder
Acronym: (Airrosti)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Majmaah University (Other)
Responsible Party: Principal Investigator, Shahnaz Hasan, PhD, Associate Professor, Majmaah University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MUREC-Oct.03/COM-2024/48
Record Dates: First submitted 2024-10-08; First posted 2024-10-16 (Actual); Last update posted 2025-05-20 (Actual); Status verified 2025-05

CONDITIONS: Rounded Shoulder Posture
Keywords: Double crossed syndrom; posture; smart phone users

STUDY DESIGN:
Intervention Model Description: Two intervention groups
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Groupe A (Active Comparator): Experimental groupe A will receive AIRROSTI exercises for 45 minutes / one session daily for five days per week.
  Interventions: Behavioral: AIRROSTI exercises
- Groupe B (Active Comparator): Group B will receive Thera band exercises for 45 minutes/one session per day for five days per week.
  Interventions: Behavioral: Thera band exercises

INTERVENTIONS:
Behavioral: AIRROSTI exercises — Group A will receive AIRROSTI exercises for 45 minutes / one session daily for five days per week
  Arms: Groupe A
Behavioral: Thera band exercises — Group B will receive Thera band exercises for 45 minutes/one session per day for five days per week.
  Arms: Groupe B

SUMMARY:
Double-crossed syndrome" refers to a specific alignment of overactive and underactive muscles in the neck, chest, and shoulders. AIRROSTI stands for Applied Integration for the Rapid Recovery of Soft Tissue Injuries. This study aims to evaluate the effectiveness of Airrosti exercises combined with TheraBand exercises in reducing pain and disability in the neck and shoulders. TheraBand exercise programs are commonly used to improve muscle activation. However, research on the effectiveness of AIRROSTI combined with TheraBand exercises for treating Double-Crossed Syndrome among smartphone users is limited, and more evidence is needed to support their effectiveness.

DETAILED DESCRIPTION:
Research objective is to evaluate the effectiveness of Airrosti and Theraband exercises in reducing pain and disability among smartphone users with Double-Crossed Syndrome. To evaluate the combined effect of Airrosti and Theraband exercises in reducing pain and disability among smartphone users with Double-Crossed Syndrome. To compare the effect of Airrosti and Theraband exercises in reducing pain and disability among smartphone users with Double-Crossed Syndrome.

ELIGIBILITY:
Inclusion Criteria:

young female participants with rounded shoulder postures. Participants aged between 18 and 25 years. No history of shoulder trauma, current shoulder pathology, thoracic scoliosis, and kyphosis deformity.

Exclusion Criteria:

Participants excluded if they received any other form of medical treatment or have thoracic scoliosis or kyphosis deformity.

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female with rounded shoulder posture
Enrollment: 60 (Estimated)
Dates: Start 2024-12-10 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
University of California at Los Angeles Activity Scale | 6 week
  Pre and post intervention measurement will be taken using University of California at Los Angeles Activity Scale. The minimum score is zero indicating several functional impairments and maximum score is 35 , indicating a normal upper limb activity.

OTHER OUTCOMES:
Double Square Test | 6week
  Pre and post intervention measurement will be taken on Double Square Test.The minimum score is 0, and the maximum score is 10, corresponding to severe disability and optimal function, respectively.
Numeric Pain rating scale | 6 week
  Pre and post intervention measurement will be taken on Numeric Pain rating scale. The minimum score is 0, indicating no pain, and maximum score is 10 , indicating worst pain imaginable.

CONTACTS AND LOCATIONS:
Overall Officials: Shahnaz Hasan associate Professor, PhD, Principal Investigator — Majmaah University
Locations (1):
- Majmaah University, Al Majma'ah, Alriyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No
There is no plan to share, it will be available with principal author and provided upon request.